CLINICAL TRIAL: NCT07204158
Title: Clinical Performance Evaluation of a Medical Device Based on Isotonic Seawater and Hyaluronic Acid Used as a Nasal Spray in Children and Adults With Nasal Dryness: a Prospective, Multicentric, Non-randomized Study in Real-life Conditions.
Brief Title: Evaluation of a Medical Device Based on Isotonic Seawater and Hyaluronic Acid Used as a Nasal Spray
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YSLab (Industry)
Collaborators: Eclevar Medtech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00666-43
Record Dates: First submitted 2025-09-22; First posted 2025-10-02 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Nasal Dryness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subject using the device (Experimental)
  Interventions: Device: Spray pompe nasal confort

INTERVENTIONS:
Device: Spray pompe nasal confort — Seawater solution with hyaluronan

SUMMARY:
The purpose of this study is to see whether the nasal spray can help improve hydration of the nasal mucosa, reduce discomfort linked to nasal dryness, and confirm its safety in patients suffering from nasal dryness.

ELIGIBILITY:
Inclusion Criteria:

* IC1. Male, female over 6 years old.
* IC2 Rhinoscopy score of at least 6, with a dryness symptom score of at least 2.
* IC3. Have a smartphone that can use MILO application, for any patient that wishes to answer the questionnaires on their phone.
* IC4. Patient and/or parent/legal guardian can understand and comply with protocol requirements and instructions.
* IC5. Patient willing to not change their daily habits including but not limited to Smoking, use of fireplace candles, air conditioning, cold air, medication and dehumidifier.
* IC6. Signed informed consent (by patient and/or parent/legal guardian).

Exclusion Criteria:

* EC1. Patients taking anticoagulants, over-the-counter or prescription systemic/topical corticosteroids, antibiotics, antihistamines, non-steroidal anti-inflammatory drugs (NSAIDs), leukotriene antagonists, topical or systemic decongestants or any treatment for relieve of nasal symptoms (except acetaminophen) in the two weeks prior to Visit 1 and during the study;
* EC2. Patient with known hyper sensibility to the study treatment;
* EC3. Patients using other nasal sprays, nasal pumps, nasal irrigation/washing devices or nasal oils, creams or gels in the two weeks prior to Visit 1 and during the study;
* EC4. Patients with any dermatological, respiratory or medical condition (e.g., asthma, pneumonia, laryngotracheobronchitis, sinusitis, nasal polyposis and chronic sinusitis, urticaria or eczema) that, in the opinion of the principal investigator, could interfere with the interpretation of study results;
* EC5. Patients with a positive medical history of any significant illness in the 2 weeks preceding the study, which, in the opinion of the principal investigator, could interfere with the interpretation of study results;
* EC6. Patients with nasal anatomical anomalies, e.g., severely deviated septum, congenital cleft lip/palate, nasal hemorrhagic diathesis (assessed by principal investigator);
* EC7. Patient that uses cocaine or other inhaled drugs
* EC8. Patients with any clinically significant co-morbid condition that, in the opinion of the principal investigator, could interfere with the interpretation of study results;
* EC9. Enrolled in another clinical trial or being in a period of exclusion from a previous clinical trial;
* EC10. Women of childbearing age (except menopausal, hysterectomized, and sterilized) are not using effective contraception (oral contraceptives, intra-uterine devices, contraceptive implants, or condoms);
* EC11. A person belonging to a population referred to in articles 64 (incapacitated subjects), 66 (pregnant or breastfeeding women), 67 (persons performing mandatory military service, persons deprived of liberty, persons who, due to a judicial decision) and 68 (patients in an emergency) of the MDR 2017/745.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-10-07 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement of the nasal dryness symptoms | From enrollment to the end of treatment at 1 week
  The changes between the baseline and day 7 in the rhinoscopy score will be assessed. The rhinoscopy score is constituted by the sum of the following symptom: dryness, atrophy, redness, oedema of the nasal mucosa and crusting. The clinician will assess each symptom on an ordinal scale of 0-4 (0 = none, 1 = mild, 2 = moderate, 3 = strong, 4 = very strong).

SECONDARY OUTCOMES:
Improvement of the total perceive Nasal symptom relief | From enrollment to the end of treatment at 1 week
  The changes between the baseline and day 7 will be assessed using the Rhinitis Sicca Symptom Score (RSSS). The RSSS is constituted by the sum of the following individual symptoms: sensation of dry nose, impairment of nasal breathing/nasal obstruction, crusting, itching/sneezing attacks, pain in the nose, anterior nasal discharge /runny nose, thick nasal discharge, desire to clear one's throat/ dry throat, impairment of smell and impairment of sleep. Patients assessed with each of these symptoms on an ordinal scale of 0-4 (0 = none, 1 = mild, 2 = moderate, 3 = strong, 4 = very strong).
Safety endpoint | From enrollment to the end of treatment at 1 week
  Adverse events, if any, will be tabulated by the investigator